CLINICAL TRIAL: NCT06463223
Title: Imaging-based Biomarkers for Liver Disease in Children With Obesity-a Longitudinal Study
Brief Title: HIBOC = Hepatic Imaging Biomarkers in Obese Children
Status: Not yet recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Hannah Hebelka, MD, Associate Professor, Sahlgrenska University Hospital
Other Study IDs: 2024-02255-01
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Elastography; Shear Wave Elastography; Shear Wave Dispersion; Attenuation Imaging; Child Obesity; Metabolic Disease; Metabolic and Genetic Disorder Affecting the Liver; Fibrosis, Liver; Diagnosis; Inflammation; Liver; Steatosis
MeSH Terms: conditions — Pediatric Obesity; Metabolic Diseases; Liver Cirrhosis; Disease; Hepatitis; Fatty Liver

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this prospective, diagnostic observational study is to learn about how imaging based markers for components of liver disease appear in children with obesity. It aims to determine whether the imaging markers (ultrasound and MRI) for liver disease can be tools to improve diagnostics for liver affection in children with obesity and to ascertain how the markers are related to multiple clinical measures, for example BMI and serology measure, and treatment effects over time.

DETAILED DESCRIPTION:
Background Childhood obesity is a global health problem with a prevalence of 10%. Overweight and obesity are strongly associated with metabolic-associated fatty liver disease (MASLD), which includes a continuum of fatty liver, hepatitis, fibrosis, and cancer. Early diagnosis is crucial for reducing morbidity and mortality but requires detailed characterization of the liver, for which invasive biopsies are the gold standard.

New ultrasound-based markers are promising, non-invasive methods for liver characterization; Shear Wave Dispersion (SWD), Shear Wave Elastography (SWE), and Attenuation Imaging (ATI) have been reported as promising for reflecting inflammation, fibrosis, and steatosis in the liver, respectively. Clinical studies are needed to validate the usefulness of these markers, particularly in children.

Purpose The study aims to determine whether imaging markers (ultrasound and MRI) for liver disease can be tools to improve diagnostics for liver affection in children with obesity and to ascertain how the markers are related to multiple clinical measures, for example BMI and serology measures, and treatment effects over time.

Material & Method This study is a prospective diagnostic observational study, including children (approximately 300) referred for obesity to several Pediatric Clinics in Västra Götaland, Sweden. Inclusion criteria are: age 9-14 years, BMI > 29, obesity > 1 year. Exclusion criteria: comorbidity that can affect the liver. Ultrasound with measurements of the livermarkers SWE, SWD, and ATI will be performed at inclusion and during annual visits over 3 years. SWE, SWD, and ATI will be compared with parameters included in clinical monitoring, such as weight, height, BMI, blood tests, blood pressure, waist circumference, physical activity, screen habits, etc. In a subcohort, estimated 50 children, with obesity-related disease as indication for referral and treatment to Queen Silvias Childrens Hospital, additionally MRI will be performed at inclusion.

Significance Imaging-based liver markers have great potential to improve diagnostics in children with obesity by reflecting liver disease without a biopsy. If these markers can be used to early diagnose liver disease before it becomes manifest, it is a significant gain. Additionally, if it is possible to distinguish between different pathoanatomical phenotypes (fibrosis/inflammation/steatosis) without a biopsy, it is possible to monitor the disease more rigorously, which opens new opportunities to optimize treatment for the individual child.

ELIGIBILITY:
Inclusion Criteria:

* Age 9 to 14 years
* New referral/first visit or follow-up annual visit at each healthcare center (Child and adolescent oriented centers) included
* BMI 30 or more
* Obesity >1 year at inclusion

Exclusion Criteria:

* Difficulty understanding written/oral information
* Comorbidities that can affect the liver (e.g., medications or diseases with known liver impact)
* Claustrophobia (applies to the MRI cohort)
* Implants or other factors that prevent MRI (applies to the MRI cohort)

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Prospectively, children referred for obesity to one of several Pediatric and Youth Clinics in the Västra Götaland region will be included. Inclusion in the study will occur via the respective clinic according to the following criteria: age 9 to 14 years, new visit or follow-up annual visit at the respective clinic, BMI of 30 or more, obesity for more than 1 year at the time of inclusion. Exclusion criteria include: difficulties in understanding written/oral information, comorbidity that can affect the liver (e.g., medications or diseases with known liver impact), claustrophobia (applies to the MRI cohort), implants or other factors that prevent MRI (applies to the MRI cohort).
  We aim to include 300 children
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Attenuation imaging | baseline, 1 year, 2 years and 3 years follow up
  an ultrasound based measure of steatosis in the liver
Shear wave dispersion | baseline, 1 year, 2 years and 3 years follow up
  an ultrasound based estimation of increased liver viscosity, seen in for example inflammation
shear wave dispersion | baseline, 1 year, 2 years and 3 years follow up
  an ultrasound based measure of liver stiffness as a reflection of liver fibrosis

SECONDARY OUTCOMES:
Magnetic Resonance Imaging fat fraction | baseline, 1 year, 2 years and 3 years follow up
  Estimation of fat content in the liver
Magnetic Resonance Imaging elastography | Baseline, 1 year,2 years and 3 years follow up
  measurement of liver stiffnes on MRI
Magnetic Resonance Imaging diffusionbased imaging | baseline, 1 year, 2 years and 3 years follow up
  Quantitative estimation of viscoelastic tissue properties
Magnetic Resonance Imaging relaxometry | Baseline, 1 year,2 years and 3 years follow up
  Detailed tissue characterization with measurement of fibrosis in the liver

OTHER OUTCOMES:
serology measures | baseline, 1 year, 2 years and 3 years follow up
  blood work
BMI | baseline, 1 year, 2 years and 3 years follow up
  body mass index